CLINICAL TRIAL: NCT02050256
Title: Improving End-of-life Care by Continuing Medical Education and Electronic Decision Making Support for General Practitioners in Denmark - an Intervention Study
Brief Title: Improving End-of-life Care by Continuing Medical Education and Electronic Decision Making Support for General Practitioners
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: due to organisational changes
Sponsor: University of Aarhus (Other)
Collaborators: Danish Cancer Society (Other); TrygFonden, Denmark (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2006802748
Record Dates: First submitted 2013-12-18; First posted 2014-01-30 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Chronic Obstructive Pulmonary Disease; Metastatic Cancer
Keywords: Palliative care; Continuing medical education; General practitioner; Electronic decision support
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Neoplasm Metastasis | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- general practioner (Other)
  Interventions: Other: continuing medical education and electronic decision support; Other: education and electronic support

INTERVENTIONS:
Other: continuing medical education and electronic decision support
Other: education and electronic support — Continuing medical education and electronic decision support to General Practitioners.

SUMMARY:
Background: Optimizing the basic palliative care has been shown beneficial to patients in end-of-life care, the general practitioner (GP) having a pivotal role in the health care system, providing comprehensive and continued medical care.

The aim of the study is to investigate the effect of a complex intervention in general practice on GPs' awareness of and confidence in providing end-of-life care.

Method: A follow-up study among 404 general practices in Central Denmark Region. The participating general practices will get the opportunity to receive education in palliative care and access to an electronic support, which provides advice on palliative care and an overview of the palliative population in each medical practice. The education and the support will focus on patients suffering from either metastatic cancer or chronic obstructive pulmonary disease (GOLD stage 4).

The end-of-life care delivered by the GPs to their deceased patients will be analysed, based on questionnaires to GPs and register data related to the deceased patients before and after the intervention, .

Primary outcomes: Place of death of deceased patients, time spent at home, and number of hospital admissions in the last three months of the patients' lives.

Secondary outcomes: Number and kinds of contacts between GPs and patients, use of relevant medicine and of the 'Safety Box'. Finally GPs' confidence concerning palliative care will be assessed in questionnaires.

ELIGIBILITY:
Inclusion Criteria:

Working as General Practitioner in the Central Region of Denmark in 2013 and onwards

-

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Place of death of deceased patients | 1 year
  Looking at the proportion of General practitioners patients dying at home in the year following the continuing medical education meeting
time spent at home the last three months of the deceased patients lives | 3 months
  Looking at all the deceased patients in one year following the continuing medical education meeting
Numbers of hospital admission the last three months of the deceased patients lives | 3 months
  Looking at all the deceased patients in one year following the continuing medical education meeting

SECONDARY OUTCOMES:
and kinds of contacts between GPs and patients in the last three months of the deceased patients lives | three months
use of relevant medicine and of the 'Safety Box' in the last three months of the deceased patients lives | three months
GPs' confidence concerning palliative care | 14 months
  assessed using questionnaire before and after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Anders B. Mr Jensen, Professor, Principal Investigator — Department of Oncology, Aarhus University Hospital, Denmark
Locations (1):
- Aarhus University, Aarhus, Denmark

REFERENCES:
- [Derived] Winthereik AK, Neergaard MA, Jensen AB, Vedsted P. Development, modelling, and pilot testing of a complex intervention to support end-of-life care provided by Danish general practitioners. BMC Fam Pract. 2018 Jun 20;19(1):91. doi: 10.1186/s12875-018-0774-x. PMID 29925332